CLINICAL TRIAL: NCT00038077
Title: Reversal of Ventricular Remodeling With Toprol-XL
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Allocation: Randomized | Masking: Double | Purpose: Treatment
Other Study IDs: 276; USMET0002
Record Dates: First submitted 2002-05-28; First posted 2002-05-29 (Estimated); Last update posted 2010-11-19 (Estimated); Status verified 2010-11

CONDITIONS: Heart Failure, Congestive
MeSH Terms: conditions — Heart Failure | interventions — Metoprolol

INTERVENTIONS:
Drug: Seloken ZOK/Toprol-XL — 50 mg
  Other Names: Toprol-XL
Drug: Seloken ZOK/Toprol-XL — 200 mg
  Other Names: Toprol-XL
Drug: Placebo

SUMMARY:
The purpose of this study is to determine whether treatment with Toprol-XL for 12 months in asymptomatic heart failure subjects will improve their heart structure and thus prevent the progression to symptomatic disease.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of stable asymptomatic heart failure.
* Documented ejection fraction less than 0.40.
* Must be able to comply with all study procedures.

Exclusion Criteria:

* Taken B-blocker therapy for longer than 1 week within 6 months prior to randomization.
* Have heart problems that would not allow B-blocker therapy.
* Receiving B-blockers therapy for any medical reason including topical B-blockers that might cause systemic absorption (e.g., glaucoma).
* Undergone certain heart surgeries, such as, prior heart transplant or cardiomyoplasty.
* Have certain heart diseases.
* Pregnant or breast feeding.
* Unlikely to survive.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300
Dates: Start 2001-08; Primary Completion 2003-09 (Actual); Study Completion 2003-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (44):
- United States (44):
  - Birmingham, Alabama
  - Mobile, Alabama
  - Little Rock, Arkansas
  - Los Angeles, California
  - Northridge, California
  - Redondo Beach, California
  - Riverside, California
  - Research Site, Farmington, Connecticut
  - Clearwater, Florida
  - Melbourne, Florida
  - Vero Beach, Florida
  - Augusta, Georgia
  - Indianapolis, Indiana
  - Jeffersonville, Indiana
  - Edgewood, Kentucky
  - New Orleans, Louisiana
  - Shreveport, Louisiana
  - Auburn, Maine
  - Baltimore, Maryland
  - Salisbury, Maryland
  - Boston, Massachusetts
  - Saint Charles, Missouri
  - St Louis, Missouri
  - Omaha, Nebraska
  - Albuquerque, New Mexico
  - Buffalo, New York
  - East Syracuse, New York
  - New York, New York
  - Rochester, New York
  - The Bronx, New York
  - Williamsville, New York
  - Burlington, North Carolina
  - Columbus, Ohio
  - Oklahoma City, Oklahoma
  - Flourtown, Pennsylvania
  - Philadelphia, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Lincoln, Rhode Island
  - Wakefield, Rhode Island
  - Tyler, Texas
  - Salt Lake City, Utah
  - Chesapeake, Virginia
  - Roanoke, Virginia
  - Green Bay, Wisconsin

REFERENCES:
- [Derived] Colucci WS, Kolias TJ, Adams KF, Armstrong WF, Ghali JK, Gottlieb SS, Greenberg B, Klibaner MI, Kukin ML, Sugg JE; REVERT Study Group. Metoprolol reverses left ventricular remodeling in patients with asymptomatic systolic dysfunction: the REversal of VEntricular Remodeling with Toprol-XL (REVERT) trial. Circulation. 2007 Jul 3;116(1):49-56. doi: 10.1161/CIRCULATIONAHA.106.666016. Epub 2007 Jun 18. PMID 17576868